CLINICAL TRIAL: NCT06915168
Title: CIPN Decision Aid to Improve Neurotoxic Chemotherapy Decision Making
Brief Title: CIPN Decision Aid for the Improvement of Chemotherapy Decision Making in Patients With Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HUM00261498; NCI-2024-10529 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HUM00261498 (Other: University of Michigan Comprehensive Cancer Center)
Record Dates: First submitted 2025-03-11; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (CIPN DecisionAid) (Experimental): Patients receive the CIPN DecisionAid on study.
  Interventions: Other: Informational Intervention; Other: Survey Administration

INTERVENTIONS:
Other: Informational Intervention — Given CIPN DecisionAid
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial studies how well a chemotherapy-induced peripheral neuropathy (CIPN) decision aid works in improving chemotherapy decision making among patients with breast cancer. CIPN involves numbness or tingling in the hands or feet and is a debilitating side effect of several commonly used classes of cancer drugs. CIPN symptoms are typically minor at first but can progress with continued treatment to severe symptoms that can affect long-term function, falls risk, and quality of life. Symptoms sometimes resolve after treatment but in patients who experienced CIPN, symptoms are still present 1 year post-treatment in about two-thirds of patients and 3 years post-treatment in approximately half of the patients. Previous studies indicate patients lack awareness of long-term CIPN symptoms. A decision aid that provides information about permanent CIPN, that helps patients understand their treatment priorities, and prepares them for a discussion with their medical oncologist may lead to improvements in treatment decision making, satisfaction with decision making, and ultimately increase patient's achievement of their treatment goals.

ELIGIBILITY:
Inclusion Criteria:

* Patients with breast cancer
* Currently receiving cycle three of taxane treatment
* Approval of medical oncologist to enroll patient
* Experiencing any CIPN based on enrollment screening question, "In the last 7 days, what was the severity of your numbness or tingling in your hands or feet at its worst? None, Mild, Moderate, Severe, Very Severe. Patient is eligible if their answer is anything except "None"
* Access to a smartphone or similar device that can complete CIPN DecisionAid via Qualtrics while in the waiting room

Exclusion Criteria:

* Inability to read or speak English

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in decision preparedness | up to 12 weeks
  Will be assessed using Question #2 on the Awareness, Preparedness, and Confidence Survey.

SECONDARY OUTCOMES:
Change in decision preparedness | up to 12 weeks
  Will be assessed using Question #2 on the Awareness, Preparedness, and Confidence Survey. A secondary analysis will be conducted using linear regression adjusting for the treatment (adjuvant versus [vs]. metastatic, paclitaxel vs. docetaxel, weekly vs. 3-weekly) and other baseline variables (e.g., age, chemotherapy-induced peripheral neuropathy [CIPN] severity).
Change in awareness | up to 12 weeks
  Will be assessed using Question #1 on the Awareness, Preparedness, and Confidence Survey.
Change in discussion confidence | up to 12 weeks
  Will be assessed using Question #3 on the Awareness, Preparedness, and Confidence Survey.
Change in decision preparedness | up to 12 weeks
  Will be assessed using Question #4 on the Awareness, Preparedness, and Confidence Survey.
Change in decision empowerment | up to 12 weeks
  Will be assessed using Question #5 on the Awareness, Preparedness, and Confidence Survey.
Discussion satisfaction | up to 12 weeks
  Will be assessed using Question #6 on the Satisfaction and Helpfulness Survey.
Decision satisfaction | up to 12 weeks
  Will be assessed using Question #7 on the Satisfaction and Helpfulness Survey.
Helpfulness | up to 12 weeks
  Will be assessed using Question #8 on the Satisfaction and Helpfulness Survey.
Taxane chemotherapy treatment decision | up to 12 weeks
  Will be assessed using Question #9 on the Satisfaction and Helpfulness Survey.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel L Hertz, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States